CLINICAL TRIAL: NCT05288036
Title: Effectiveness of Proprioceptive Neuromuscular Facilitation for Improving for Shoulder Biomechanical Parameters, Function, and Pain After Axillary Lymph Node Dissection: a Randomized Controlled Study
Brief Title: Effectiveness of PNF Training for Improving for Muscle Strength, Function, and Pain After Axillary Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.184
Record Dates: First submitted 2021-12-26; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Muscle Strength
Keywords: Proprioceptive Neuromuscular Facilitation; Pain; Axillary Disease
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioceptive Neuromuscular Rehabilitation group (Experimental): PNF techniques; It is based on facilitating the responses of neuromuscular mechanisms by stimulating proprioceptors. It is a method used to improve active movement ability by increasing muscle strength, to increase muscle endurance, to improve stabilization at the point where the technique is applied within the movement pattern.
  Interventions: Other: Proprioceptive Neuromuscular Rehabilitation group
- Progressive Resistance Exercise Group (Experimental): Progressive resistance training (PRT) is a method for increasing muscle strength and endurance based on the determination of the amount of resistance appropriate for the individual. Free weights and resistance machines are used in the practice of this technique.To facilitate continued adaptation, training intensity (i.e. load) and training volume (i.e. number of sets) are progressively increased, and exercises are adjusted as indicated throughout the training regimen, to attenuate the onset of a plateau in physiological adaptation.
  Interventions: Other: Progressive Resistance Exercise Group
- Control Group (Active Comparator): This group was created to determine the amount of self-healing of the disease in the process. The approach was taken in a way that did not affect the outcome measures.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Rehabilitation group — The PNF technique was performed in the supine position with the hip joints of the patients in 30° flexion and the lower extremities in semi-flexion. The application was performed in 2 different diagonal and 4 different patterns (flexion-abduction-external rotation/extension-abduction-internal rotation, and flexion-adduction-external rotation/extension-abduction-internal rotation) of the upper extremity. When starting the exercise, the muscles were first brought to their longest position and the patient was asked to move in the direction of the pattern with resistance (concentric contraction) and to maintain this position for 6 seconds at the end of the pattern (isometric contraction). Then, while the therapist was taking the patient's arm to the starting position, the patient was asked to prevent movement (eccentric contraction). All of these moves counted as one repetition. 3 sets of 8-12 repetitions were performed for each pattern.
  Other Names: PNF
  Arms: Proprioceptive Neuromuscular Rehabilitation group
Other: Progressive Resistance Exercise Group — Strengthening exercises targeting the upper extremity main muscles were applied to the PRE group with progressive resistance. Dumbbells and sandbags were used as resistance equipment. resistance intensity; 50-80% of a repetition maximum (RM) was determined according to the patient's tolerance. The exercises were applied as 8-12 repetitions and 3 sets. A rest period of 60-90 seconds was allowed between each set. After the 4th week of the training, 1 RM was measured again and the resistance density was updated. The 8 strengthening exercises to be applied were created by taking examples from the literature and in accordance with the "Guidelines for implementing exercise programs exercise programs for cancer patients". These exercises are: "dumbbell fly", "triceps extension", "biceps curl up", "one-arm bent over row", "dumbbell sides rise", "lifting the arm forward", "wrist curl" and side lying shoulder internal -external rotation".
  Other Names: PRE
  Arms: Progressive Resistance Exercise Group
Other: Control Group — The patients in the control group were instructed to continue their usual daily lives (not changing their physical activity levels, diet, drug use, etc.) until the date of re-evaluation after the initial evaluation. Information was given about the upper extremity normal range of motion exercises that they could apply at home, and a brochure was given.
  Arms: Control Group

SUMMARY:
Breast cancer is the most common type of cancer affecting women of all ages worldwide. Advanced and comprehensive treatment options have increased survival rate and life expectancy, necessitating a focus on the complications of breast cancer treatment. Although axillary lymph node dissection (ALND) causes high morbidity, it is an integral part of surgical treatment in patients with invasive breast cancer and axillary lymph node metastasis. Axillary lymph node dissection and radiotherapy are associated with pain, physical symptoms, and decreased functional abilities in the upper extremity. This study aimed to compare the potential effects of proprioceptive neuromuscular facilitation (PNF) technique on muscle strength, pain and functionality in this patient group with progressive resistance exercise (PRT).

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer affecting women of all ages worldwide. An increase in the incidence of breast cancer is observed with the effect of widespread screening programs today. Improved and comprehensive treatment options (surgery, radiotherapy, systemic adjuvant and neoadjuvant therapy, hormonal therapy) have increased the survival rate and life expectancy. This has necessitated a focus on the short, medium and long term complications of breast cancer treatment and their management.

Although axillary lymph node dissection (ALND) causes high morbidity, it is an integral part of surgical treatment in patients with invasive breast cancer and axillary lymph node metastasis (2). Radiotherapy is routinely used to reduce the local recurrence rate after ALND. 73% of the patients who received these treatments reported that they had at least 1 complaint of limitation of shoulder joint range of motion, loss of strength in the operated arm, pain, lymphedema numbness, fibrosis, fatigue, and inability in activities of daily living in the postoperative period.

It is known that the muscle strength of the operated side arm is less than the strength of the contralateral extremity and the strength of healthy women due to many reasons such as deterioration of the soft tissue integrity of the chest wall with surgery, inactivity tendencies of the patients due to protecting the operated arm, adhesions that may occur with radiotherapy, and fibrosis formations making movement difficult. In addition, one-third of women with breast cancer treated with surgery experience permanent loss of strength in their upper extremity muscles for more than 1 year after treatment. According to the results of a study investigating the causes of persistent pain after breast cancer treatment, ALND and radiotherapy administration are the two main risk factors for persistent pain, and 21% of women who have ALND experience persistent shoulder/arm pain throughout their lives. Adequate muscle strength and no pain during movement are of great importance for the quality of movement and for the smooth performance of daily life activities. In a study on patients' evaluation of their own upper extremity functionality, women receiving breast cancer treatment stated that they were more functionally limited than their healthy peers and had difficulties in activities of daily living. In a study of large populations, it was reported that the prevalence of functional limitations in women receiving breast cancer treatment ranged from 18% to 54%. Functional limitations complicate the situation and bring the need for additional treatments to improve daily living activities, as well as the application of treatments related to the current disease to the patient.

Exercise is one of the most commonly used modalities in the rehabilitation of patients receiving breast cancer treatment. The main goals of exercise in these patients are to increase muscle strength, reduce pain, increase limited range of motion and contribute to the ability to continue activities of daily living. Resistance exercises are the most commonly used method to provide strength gain and restoration, and there are many studies in the literature on their positive effects on strength enhancement in the affected extremity.

The proprioceptive neuromuscular facilitation (PNF) technique applied for the treatment of the operated shoulder/arm may play a role in regaining strength, power and endurance by increasing the response of neuromuscular mechanisms by stimulating the proprioceptors. At the same time, there are studies showing that this treatment modality provides a significant reduction in shoulder-arm pain and provides painless quality movement. With this technique, functional restoration is provided thanks to the movement patterns applied in the diagonal direction. These gains reveal the importance of using the PNF technique more frequently in breast cancer patient groups where it is applicable.

The PNF technique is emerging as a therapeutic option to increase muscle strength, reduce pain, and improve functionality in patients treated for breast cancer with ALND. The aim of this study is to compare the efficacy of resistance exercise and PNF technique, the effectiveness of which was defined on the patient, on the aforementioned subjects.Patients who applied to Istanbul Medipol University General Surgery Department for routine control after breast cancer treatment were determined. Individuals who were willing to participate and met the inclusion criteria were divided into 3 groups (PNF, progressive resistant ex., control) using the website www.randomizer.org.

Exercise was applied to both Proprioceptive Neuromuscular Facilitation (PNF) and Progressive Resistance Exercise (PRE) groups, 2 days a week for 8 weeks. Each session lasted an average of 1 hour. Exercise sessions; It was carried out under the supervision of the same physiotherapist with experience in the field and individually with each patient. At the beginning and at the end of the treatment, warm-up-cooling exercises including mild stretching exercises to increase the range of motion were performed for 5-10 minutes. In both groups, exercises were performed only for the affected extremity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with stage II-III breast cancer
* 30-65 years old
* ALND was performed by the same surgeon regardless of breast resection level.
* Receiving radiotherapy
* Individuals who spent the first six months after surgery were included in the study.

Exclusion Criteria:

* Diagnosed with stage IV or metastatic breast cancer
* Developing bilateral breast cancer
* Developing lymphedema in the postoperative period
* Any contraindication to exercise
* Participating in any physiotherapy program for the upper extremity in the last 6 months
* Have significant cardiac, pulmonary or metabolic comorbid disease
* Individuals with communication problems were excluded from the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients were included in the study.
Enrollment: 66 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Isokinetic dynamometer | "8 weeks"."Two measurements were made to evaluate the change before treatment (baseline) and at the end of treatment (8 weeks later).".
  Humac Norm, model 770, Computer Sports Medicine Inc., Stoughton, USA was used to biomechanically evaluate shoulder flexors/extensors, abductor/adductors, internal/external rotators. Muscle strength was measured at 60°/s, muscle strength at 120°/s, endurance at 180°/s angular velocity and in concentric/concentric mode. 5 repetitions at 60°/s and 120°/s angular velocity, and 15 repetitions at 180°/s angular velocity were performed at the measured active range of motion. The measurement was performed only on the operated side upper extremity. A rest period of 2 minutes was provided between series of each muscle group and 5 rest periods between different movement patterns. For each angular velocity, the first trial was subtracted, and the average peak torque value of the remaining repetitions (the force produced by the individuals at the maximum during the angular velocity) was recorded in Newton-meters (Nm).
Disabilities of the Arm, Shoulder, and Hand (DASH) | "8 weeks"."Two measurements were made to evaluate the change before treatment (baseline) and at the end of treatment (8 weeks later).".
  The scale includes 30 questions about symptoms (5 items) and functionality (25 items). In this study, business/sport-specific additional modules of the scale were not used. Each item offers 5 answer options and is scored on a likert scale from 1 to 5. 1: reflects 'no difficulty' and 5: reflects 'serious difficulties'. The resulting scores for all items are then used to calculate the total score from 0 (no disability) to 100 (most severe disability) (16). It is accepted as the most consistent test in terms of construct validity and responsiveness in examining upper extremity problems in individuals undergoing breast cancer treatment.
Visual Analogue Scale (VAS) | "8 weeks". "Two measurements were made to evaluate the change before treatment (baseline) and at the end of treatment (8 weeks later).".
  The patients were asked to mark their pain levels in the breast, shoulder and axilla regions on the affected side during rest and activities of daily living on a 10 cm scale (0=no pain, 10=worst pain ever experienced). The distance (cm) between the zero point and the point marked by the patient indicates the level of pain.
Global Rating Of Change Scale (GRC) | "8 weeks". "Baseline and 8th week".
  The Global Rating of Change Scale (GRC) contains a single question in which the patient can rate how much he has improved retrospectively from his own perspective. The validity and reliability of the GRC scale has been verified and is widely used in the assessment of change for musculoskeletal problems. 7 different answers (-3: much worse, 2: worse, -1: slightly worse, 0: the same, 1: a little better, 2: quite good, 3 They were asked to answer by choosing one of the :much better) options. In scoring, scoring can be done according to a 7-point Likert evaluation, as well as calculations can be made using negative scores. This scale was applied only to the study groups in the post-treatment measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Basim, Assoc. prof., Study Director — Medipol University
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Hindle KB, Whitcomb TJ, Briggs WO, Hong J. Proprioceptive Neuromuscular Facilitation (PNF): Its Mechanisms and Effects on Range of Motion and Muscular Function. J Hum Kinet. 2012 Mar;31:105-13. doi: 10.2478/v10078-012-0011-y. Epub 2012 Apr 3. PMID 23487249
- [Background] da Silveira DSP, Dos Santos MJ, da Silva ET, Sarri AJ, das Neves LMS, Guirro ECO. Proprioceptive neuromuscular facilitation in the functionality and lymphatic circulation of the upper limb of women undergoing breast cancer treatment. Clin Biomech (Bristol). 2020 Dec;80:105158. doi: 10.1016/j.clinbiomech.2020.105158. Epub 2020 Aug 31. PMID 32896753
- [Background] Kraemer WJ, Ratamess NA. Fundamentals of resistance training: progression and exercise prescription. Med Sci Sports Exerc. 2004 Apr;36(4):674-88. doi: 10.1249/01.mss.0000121945.36635.61. PMID 15064596
- [Background] Cormie P, Singh B, Hayes S, Peake JM, Galvao DA, Taaffe DR, Spry N, Nosaka K, Cornish B, Schmitz KH, Newton RU. Acute Inflammatory Response to Low-, Moderate-, and High-Load Resistance Exercise in Women With Breast Cancer-Related Lymphedema. Integr Cancer Ther. 2016 Sep;15(3):308-17. doi: 10.1177/1534735415617283. Epub 2015 Nov 17. PMID 26582633
- [Derived] Guloglu S, Basim P, Algun ZC. Efficacy of proprioceptive neuromuscular facilitation in improving shoulder biomechanical parameters, functionality, and pain after axillary lymph node dissection for breast cancer: A randomized controlled study. Complement Ther Clin Pract. 2023 Feb;50:101692. doi: 10.1016/j.ctcp.2022.101692. Epub 2022 Nov 11. PMID 36528984

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT05288036/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT05288036/ICF_001.pdf